CLINICAL TRIAL: NCT05435378
Title: Effect of Adjunctive Use of Vitamin B3 and B9 on Myeloperoxidase Level in the GCF of Patients With Stage I and II Periodontitis, a Randomized, Parallel Group, Double Blinded, Placebo Controlled Study
Brief Title: Effect of Adjunctive Use of Vitamin B3 and B9 on Myeloperoxidase Level in the GCF of Patients With Stage I and II Periodontitis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Elham Essam Hussien Elkholy, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PER 3.3.2
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Periodontitis Stage I; Periodontal Diseases; Periodontal Inflammation; Periodontal Attachment Loss; Periodontitis; Periodontitis Stage II
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Periodontal Attachment Loss | interventions — Niacinamide; Tablets; Niacin; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Trial medication will be dispensed in similar colored capsules, prepacked in similar opaque white plastic jars of 30 capsules each so that neither patient nor investigator (whom is also the care provider) will know whether patient was receiving vitamin B3, B9 or placebo. the outcome assessor will be given the data coded without knowing the data for the group of patients corresponding to which intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vitamin B3 (Experimental): Vitamin B-3 capsule consists of Manufacturer: DSM Nutritional products Ltd generic name: nicotine amide Constituent components: 100mg of nicotine amide Route of administration: orally dosing schedule:1capsule/day/ before meal duration: for 30 days
  Interventions: Drug: Vitamin B3 100 MG Oral Tablet; Procedure: full mouth non surgical periodontal treatment
- Vitamin B-9 (Experimental): Vitamin B-9 capsule Manufacturer: Hebei Jiheng pharmaceutical Co. Ltd generic name: folic acid. Constituent components: 5 mg of folic acid. Route of administration: orally dosing schedule: 1capsule/day/before meal duration: for 30 days
  Interventions: Drug: vitamin B9; Procedure: full mouth non surgical periodontal treatment
- Placebo capsule (Placebo Comparator): Placebo capsule Manufacturer: Shivangan Foods & Pharma Products Pvt. Ltd Constituent components: inactive fillers Route of administration: orally dosing schedule: 1capsule/day/before meal duration: for 30 days
  Interventions: Drug: Placebo; Procedure: full mouth non surgical periodontal treatment

INTERVENTIONS:
Drug: Vitamin B3 100 MG Oral Tablet — After the non surgical treatment and the oral hygiene instructions The systemically administered vitamin B3 capsules will then given to the patients under the previously mentioned dosage.
  Other Names: niacin; niacinamide; nicotinamide
  Arms: vitamin B3
Drug: vitamin B9 — After the non surgical treatment and the oral hygiene instructions the systemically administered vitamin B9 capsules will then given to the patients under the previously mentioned dosage.
  Other Names: Folic acid; Folate; folacin
  Arms: Vitamin B-9
Drug: Placebo — After the non surgical treatment and the oral hygiene instructions The systemically administered placebo capsules will then given to the patients under the previously mentioned dosage.
  Other Names: inactive drug
  Arms: Placebo capsule
Procedure: full mouth non surgical periodontal treatment — full mouth scaling and debridement will be done by the primary investigator using ultrasonic scaler and periodontal curettes. After the non surgical treatment patients will be given oral hygiene instructions where they will be instructed to brush twice daily and shown how to brush using the horizontal scraping technique they will also be instructed to use the dental floss and shown how to use it.

SUMMARY:
this study addresses the effect of the vitamin B3 and vitamin B9 on the periodontal healing at the sites of periodontal destruction due to periodontitis and evaluate its added effect to the conventional non-surgical periodontal treatment on its pivotal role in the biological activities and repair in the body in general and the periodontium in specific. The research will be conducted on patients suffering from stage I and II periodontitis that typically are to be treated with non surgical periodontal therapy, the rationale of the non surgical periodontal treatment is eliminating the plaque biofilm responsible for stimulation of host immune defense causing the inflammation and hence suppressing the periodontal destruction.

the trial is targeting enhancing the treatment effect by the administration of vitamin B3 and B9 supplements which will target the host inflammatory reaction itself and directly suppressing it as well as enhancing the periodontal regeneration and the gain of the lost attachment.

DETAILED DESCRIPTION:
This study is a parallel group randomized, Double-blinded, Placebo-controlled clinical trial The follow up of this study is set to be in a three months interval in order to monitor the effect of the periodontal treatment with/without vitamin B-3 and B-9 supplement on the periodontal repair and regeneration

The eligible patients will be randomized into three groups with four interventions:

1. Non-surgical scaling and debridement with placebo
2. Non-surgical scaling and debridement with vitamin B-3
3. Non-surgical scaling and debridement with vitamin B-9 Before intervention, a gingival cervicular fluid sample will be collected for all groups to measure the myeloperoxidase level at baseline before treatment then a full mouth scaling and debridement will be done by the primary investigator using ultrasonic scaler and periodontal curettes. After the non surgical treatment patients will be given oral hygiene instructions where they will be instructed to brush twice daily and shown how to brush using the horizontal scraping technique they will also be instructed to use the dental floss and shown how to use it. The systemically administered vitamin B or placebo capsules will then given to the patients and instructed to be taken once daily for 30 days. Patients are instructed not to take any vitamin B supplementations during the period of treatment, patients are also instructed to discontinue using the drug if any allergic reaction appeared and directly report it to the investigator.

Periodontal maintenance appointments which will include a review of medical and dental histories, supra- and subgingival instrumentation if needed, and oral hygiene instructions and motivation will be performed at 14, 30, 60 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* patients with gingivitis or stage I/II periodontits. The presence of gingivitis and the presence/severity of periodontitis is registered using the American Academy of Periodontology 2017 workshop published definition With this method, patient was identified affected by periodontits when ''Interdental CAL is detectable at ≥2 non-adjacent teeth, or Buccal/oral CAL ≥3 mm with pocketing >3 mm is detectable at ≥2 teeth'' (Toentti et al, 2018) with grade I severity being cases with interdental CAL from 1-2mm and grade II severity being cases with interdental CAL from 3-4 mm

Exclusion Criteria:

* Patients incapable of giving informed consent
* Patients unable to attend the 3-month follow-up
* Patients with interdental CAL >4mm
* Patient requiring surgical periodontal treatment
* Patients on systemically administered vitamin B or vitamin B-complex
* Patients undergoing chemo- or immunosuppressive therapy over the previous 5 years
* Patients treated or undergoing treatment with intravenous amino-bisphosphonates
* Patients with poor oral motivation
* Substance abusers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
change form the baseline in myeloperoxidase level in gingival crevicular fluid at 90 days | baseline and 90 days
  biological sample of GCF will be collected and the enzyme level in GCF will be measured using The enzyme-linked immunosorbent assay (ELISA)
change form the baseline in clinical attachment level at 90 days | baseline and 90 days
  Using a University of North Carolina probe (UNC) -15 measuring the distance from the cement-enamel junction to the base of the periodontal pocket at six sites of the tooth (mesiobuccal-distobucal-midbucal-mesiolingual-distolingual-midlingual)

SECONDARY OUTCOMES:
change form the baseline in periodontal pocket depth at 90 days | baseline and 90 days
  Using UNC15 periodontal probe measuring the distance from the gingival margin to the base of the pocket at six sites of the tooth (mesiobuccal-distobucal-midbucal-mesiolingual-distolingual-midlingual)
change form the baseline in bleeding on probing at 90 days | baseline and 90 days
  Using UNC15 periodontal probe at six sites of the tooth (mesiobuccal-distobucal-midbucal-mesiolingual-distolingual-midlingual) recorded at each site as present or absent
change form the baseline in plaque index at 90 days | parameter will be evaluated at baseline and at 90 days
  Manual UNC periodontal probe setting Scores of :
  0: No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of a disclosing solution or by using the probe on the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin, which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Patient satsification | Parameter will be evaluated at 90 days
  VAS for patient satisfaction a Scale from 1-10 0 (completely dissatisfied)to 10 (completely satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Riham Omar, professor, Study Chair — main supervisor

IPD SHARING:
Plan to Share IPD: No